CLINICAL TRIAL: NCT03977493
Title: IncobotulinumtoxinA (Xeomin) to Treat Focal Hand Dystonia: a Double-blind Placebo-controlled Randomized Multicenter Study: The "SwissHandSpasm" Study
Brief Title: IncobotulinumtoxinA (Xeomin) to Treat Focal Hand Dystonia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alain Kaelin (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Alain Kaelin, Director of the Neurocenter of Southern Switzerland, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSI-BTX-001
Record Dates: First submitted 2019-04-19; First posted 2019-06-06 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Focal Hand Dystonia
MeSH Terms: conditions — Dystonia, Focal, Task-Specific | interventions — incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xeomin® (Active Comparator): Intramuscular IncobotulinumtoxinA (Xeomin®) injection under guidance (EMG and/or sonographic monitoring), 2.5 to 40 U in each muscle (max. 5 forearm- and/or hand muscles).
  Interventions: Drug: Xeomin
- Placebo concentrate (Placebo Comparator): Intramuscular Placebo injection under guidance (EMG and/or sonographic monitoring), in each muscle (max. 5 forearm- and/or hand muscles).
  Interventions: Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: Xeomin — One injection of 2.5 to 40 U in each muscle. Injection repeated after 6 weeks if considered necessary
  Arms: Xeomin®
Drug: Placebo - Concentrate — One injection in each muscle.
  Arms: Placebo concentrate

SUMMARY:
This study is a multicenter, double-blind, randomized placebo controlled, parallel group, superiority trial in order to test the superiority of intramuscular injections of IncobotulinumtoxinA against placebo using a 1:1 allocation ratio.

DETAILED DESCRIPTION:
After a baseline evaluation, each patient will receive a first injection of IncobotulinumtoxinA or placebo (50:50 randomization) in a double blinding setting. Assessment of the Focal hand dystonia (FHD) will be done at each site by an investigator blinded to the treatment.

A first evaluation of the efficacy will be performed after 6 weeks. After 6 weeks, patients unsatisfied with treatment and wishing to continue the treatment will receive an injection of IncobotulinumtoxinA regardless of the treatment arm they were initially assigned to at baseline. These patients will subsequently be excluded from the study.

A second assessment will be performed after 12 weeks (only for patients not receiving a second injection of IncobotulinumtoxinA at week 6).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age ≥ 18 years
* Focal hand dystonia (FHD). Diagnosis must be made by a neurologist specialized in movement disorder (at least 2 years specific training, all partners listed have at least 2 years training)
* Both idiopathic and secondary FHD are allowed
* Both drug naive subjects and subjects previously treated with other BoNT-A will be included
* Patients must be willing and able to comply with the study procedures
* Female patients of childbearing potential must agree to use an effective method of contraception during the treatment period

Exclusion Criteria:

* Presence of spasticity, or other central sensorimotor lesion of motor system other than dystonia in the affected limb
* Peripheral nerve lesion (diagnosis either clinical or electrophysiological) in the affected limb, for example with a muscle weakness at baseline
* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to BoNT-A toxins including IncobotulinumtoxinA
* Doses and schedules of any ongoing treatment with potential confounding drugs such as muscle relaxants (for example Tolperison, Tizinadid, Baclofen, Mestinon, Dantrolen), benzodiazepine, neuroleptics or antidepressants have to be kept unchanged throughout the study and no changes should be made between the first trial injection and the end of study visit at week 12.
* Previous treatment with other BoNT-A less than 3 months before the inclusion in this study
* Women who are pregnant or breast feeding,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Severe depression (>29 as measured with the Beck Depression Inventory, see Appendix 8) or other relevant psychiatric disorder
* INR > 2 on the day of injection if the patient is anticoagulated. If INR > 2, the study injection will be delayed until the return to a safer INR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-02-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of IncobotulinumtoxinA on focal hand dystonia (FHD) | 6 weeks
  To evaluate patient's subjective impairment due to FHD on VAS for handwriting. The VAS for handwriting is a self-assessment scale drawn by the patients on a 10-cm line, on which 0 indicates the worst possible situation and 10 the best possible situation.

SECONDARY OUTCOMES:
Evaluation of the efficacy of IncobotulinumtoxinA on FHD | 12 weeks
  To evaluate patient's subjective impairment due to FHD on VAS for handwriting. The VAS for handwriting is a self-assessment scale drawn by the patients on a 10-cm line, on which 0 indicates the worst possible situation and 10 the best possible situation.
Evaluation of the effect of IncobotulinumtoxinA on FHD symptoms severity | 6 and 12 weeks
  To measure change in symptoms severity by using the Symptom Severity Scale (SSS). Total SSS score ranges from 10 (best possible) to 43 (worst possible).
Evaluation of the effect of IncobotulinumtoxinA on functional status | 6 and 12 weeks
  To measure change in functional status by using the Functional Status Scale (FSS). Total FSS score ranges from 0 (best possible) to 40 (worst possible).
Evaluation of the effect of IncobotulinumtoxinA on writer's cramp improvement | 6 and 12 weeks
  To measure the change in writer's cramp measured by the Writer's Cramp Rating Scale (WCRS) - only part A. Total WCRS score ranges from 0 (no improvement) to 28 (marked improvement).
Evaluation of the effect of IncobotulinumtoxinA on disease improvement | 6 and 12 weeks
  To measure the change in the physician's clinical evaluation of the disease by using the CGI-improvement scale. The CGI-improvement scale ranges from 0 to 4 (none, minimal, mild, moderate, excellent).
Evaluation of the effect of IncobotulinumtoxinA on writing pressure | 6 and 12 weeks
  To measure the change in writing pressure by using a pressure sensitive-tablet. Writing Movement pressure will be measured in Pascal.
Evaluation of the effect of IncobotulinumtoxinA on writing speed | 6 and 12 weeks
  To measure the change in writing speed by using a pressure sensitive-tablet. Writing movement speed will be measured in seconds.
Evaluation of the effect of IncobotulinumtoxinA on muscle strength | 6 and 12 weeks
  To measure the change in muscle strength by using the Medical Research Council Scale for Muscle strength. The patient's effort is graded on a scale of 0 (normal muscle) to 5 (no movement).
Evaluation of the responders to IncobotulinumtoxinA treatment | 6 and 12 weeks
  Number of patients showing an improvement of FHD by ≥ 1 points over baseline
Evaluation of the overall satisfaction of the patients following IncobotulinumtoxinA treatment | 6 weeks
  Patients will answer the following two questions: a) Considering all advantages and disadvantages of this treatment, is the improvement such that you wish to continue this treatment or not? Yes/No b) Do you think that you would need an injection of IncobotulinumtoxinA today? Yes/No
Need of re-injection | 6 weeks
  The physician will judge about whether an injection with IncobotulinumtoxinA is recommended or not (Yes/No)
Safety outcomes: adverse events | 6 and 12 weeks
  Incidence and severity of adverse reactions (mild, moderate, severe).
Safety outcomes: pain | 6 and 12 weeks
  Pain assessed by VAS scale. The VAS for pain is a self-assessment scale drawn by the patients on a 10-cm line, on which 0 indicates no pain and 10 an extreme amount of pain.
Safety outcomes: weakness | 6 and 12 weeks
  Weakness assessed by using the CGI-side effect scale and CGI-weakness scale. CGI-side effect scale ranges from 0 to 3 (no, mild, marked, severe side effects). CGI-weakness assessment scale ranges from 0 to 4 (none, <25%, 26-50%, 51-75%, 76-100% reduction in normal strength).
Evaluation of the effect of IncobotulinumtoxinA on depressive symptoms | 6 and 12 weeks
  To measure the change in depressive symptoms by using the Beck Depression Inventory (BDI). Total BDI score ranges from 0 to 63 with scores > 29 indicating severe depression and > 40 extreme depression.

CONTACTS AND LOCATIONS:
Locations (5):
- Switzerland (5):
  - Inselspital - University Hospital Berne, Bern
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne
  - Neurocentro della Svizzera Italiana, Lugano
  - Neurocenter of St. Gallen, Sankt Gallen
  - USZ- Univerity Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided